CLINICAL TRIAL: NCT02259010
Title: A Phase 1 Study to Evaluate the Effect of Itraconazole, a Strong CYP3A Inhibitor, on the Pharmacokinetics of Alisertib (MLN8237) in Adult Patients With Advanced Solid Tumors or Relapsed/Refractory Lymphoma
Brief Title: A Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of Alisertib in Participants With Advanced Solid Tumors or Relapsed/Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C14020; U1111-1161-5039 (Registry Identifier: WHO)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Advanced Solid Tumors; Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg (Experimental): All participants were to complete Part A prior to Part B. Part A: Alisertib 30 mg, tablets, orally, on Days 1 and 10 plus itraconazole, 200 mg, oral solution, once daily on Days 5 to 13. Part A and B were separated by a washout period of at least 10 days (and up to 4 weeks). Part B: Alisertib 50 mg, tablets, orally, twice daily, for 7 days in 21-day cycles until disease progression or unacceptable toxicity (up to 16 cycles).
  Interventions: Drug: Alisertib; Drug: Itraconazole

INTERVENTIONS:
Drug: Alisertib — Alisertib tablets
Drug: Itraconazole — Itraconazole oral solution
  Other Names: SPORANOX®

SUMMARY:
This study will assess the effect of multi-dose administration of itraconazole on the single-dose pharmacokinetics (PK) of alisertib.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib. Alisertib is being tested in adult participants with advanced solid tumors or relapsed refactory lymphoma. The study will look at the effect of the pharmacokinetics (how the drug moves through the body) of alisertib in the presence and absence of itraconazole.

This is an open label study. Participants will receive:

* Alisertib tablets 30 mg in Part A and 50 mg in Part B
* Itraconazole oral solution 200 mg in Part A

Participation in Part A is approximately 25 days. Part B participation is repeating 21-day cycles. The maximum duration of treatment with alisertib will be 12 months (approximately 16 cycles) unless it is determined by the investigator, with agreement by the sponsor, that a participant would derive clinical benefit from continued treatment beyond 12 months.

This multi-center study will take place in the United States.

ELIGIBILITY:
Inclusion Criteria

1. Male and female participants 18 years of age or older.
2. Participants with histologic or cytologic diagnosis of advanced or metastatic solid tumors or lymphomas for which no curative or life-prolonging therapies exist.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria

1. Systemic treatment with moderate or strong CYP3A inhibitors or inducers must be discontinued at least 14 days before the first dose of alisertib, and the use of these agents is not permitted during the study (except for the protocol-specified administration of itraconazole).
2. Known gastrointestinal (GI) abnormality (including recurrent nausea or vomiting) or GI procedure that could interfere with or modify the oral absorption or tolerance of alisertib.
3. Known hypersensitivity or intolerance to itraconazole or similar class agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2015-03-27 (Actual); Study Completion 2016-10-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - St Louis, Missouri
  - Oklahoma City, Oklahoma
  - Germantown, Tennessee
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 22 October 2014 to 21 October 2016. Data cutoff for the primary analysis was 27 March 2015.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or lymphomas were enrolled to receive alisertib 30 mg tablets, orally along with itraconazole 200 mg, oral solution in part A followed by alisertib 50 mg, tablets in part B.
Period: Overall Study
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
Started | 24
Completed | 19 (Completed=Completed protocol-specified dosing and PK assessment.)
Not Completed | 5
Not completed — Didn't Completed Dosing; PK Assessment | 5

BASELINE CHARACTERISTICS:
Population: Safety Population is defined as all participants who received at least 1 dose of any study drug and was used for all safety analyses.
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20
  Black or African American | 2
  Asian | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Height [Mean (Standard Deviation); unit: cm] | 168.3 (8.99)
Weight [Mean (Standard Deviation); unit: kg] | 85.55 (25.641)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area=square root of (height [cm]*weight [kg]/3600).
  m^2 | 1.983 (0.3024)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Concentration of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose in Cycle 1 for alisertib without itraconazole arm; Day 10 pre-dose and at multiple time points (up to 96 hours) post-dose in Cycle 1 for alisertib with itraconazole arm
Population: Pharmacokinetic (PK) -Evaluable Population included participants who completed the protocol-specified dosing at Part A and had sufficient PK assessment to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Alisertib Without Itraconazole: Alisertib 30 mg, tablets, orally, on Day 1 in Part A.
- Alisertib With Itraconazole: Itraconazole, 200 mg, oral solution, once daily on Days 5 to 13 along with alisertib 30 mg, tablets, orally, on Day 10 in Part A .
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 19 | 19
nmol/L | 1060.3 (403.90) | 1002.8 (263.81)
Statistical Analysis 1: Comparison: Alisertib Without Itraconazole vs Alisertib With Itraconazole; Test type: Superiority or Other; Least Squares Mean Ratio = 0.98, 90% CI 2-sided [0.82 to 1.19] — Estimates were obtained using a mixed effects model of log (PK parameter) with fixed terms for the itraconazole effect and random terms for participant within period

2. Primary Outcome: AUC(Last): Area Under the Plasma Concentration Curve From Time 0 to the Time of the Last Quantifiable Concentration of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: PK-Evaluable Population included participants who completed the protocol-specified dosing at Part A and had sufficient PK assessment to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 19 | 19
hr*nmol/L | 15541.6 (9119.52) | 20219.5 (9930.93)
Statistical Analysis 1: Comparison: Alisertib Without Itraconazole vs Alisertib With Itraconazole; Test type: Superiority or Other; Least Squares Mean Ratio = 1.35, 90% CI 2-sided [1.02 to 1.79] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration Curve From Time 0 to Infinity of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: PK-Evaluable Population included participants who completed the protocol-specified dosing at Part A and had sufficient PK assessment to reliably estimate PK parameters. Here number of participants analyzed are the participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 13 | 15
hr*nmol/L | 16804.6 (9232.87) | 23488.7 (13262.31)
Statistical Analysis 1: Comparison: Alisertib Without Itraconazole vs Alisertib With Itraconazole; Test type: Superiority or Other; Least Squares Mean Ratio = 1.39, 90% CI 2-sided [0.99 to 1.95] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: CL/F: Oral Clearance of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: PK-Evaluable Population included participants who completed the protocol-specified dosing at Part A and had sufficient PK assessment to reliably estimate PK parameters. Here, number of participants analyzed are the total number of participants who were evaluable to this outcome measure at specified endpoint.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 13 | 15
L/hr | 4.416 (2.4007) | 3.177 (1.5765)

5. Secondary Outcome: Tmax: Time to Reach Maximum Plasma Concentration of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 19 | 19
hr | 2.920 (2.3710) [1.07 to 10.00] | 2.920 (2.0244) [1.83 to 7.82]

6. Secondary Outcome: Terminal Phase Elimination Half-Life of Alisertib in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 13 | 15
hr | 22.55 (10.316) | 25.37 (9.215)

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Alisertib Metabolites M1 and M2 in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 18 | 19
nmol/L
  Metabolite 1 (M1): number analyzed (Participants) | 18 | 18
  Metabolite 1 (M1) | 409.4 (479.92) | 450.0 (664.65)
  Metabolite 2 (M2) | 114.0 (52.71) | 103.5 (99.28)

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib Metabolites M1 and M2 in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 18 | 19
hr
  Metabolite 1 (M1): number analyzed (Participants) | 18 | 18
  Metabolite 1 (M1) | 3.090 [1.00 to 23.10] | 3.800 [1.98 to 10.00]
  Metabolite 2 (M2) | 9.360 [2.95 to 47.70] | 23.600 [5.73 to 95.30]

9. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib Metabolites M1 and M2 in Presence and Absence of Itraconazole in Part A
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | Alisertib Without Itraconazole | Alisertib With Itraconazole
Number analyzed (Participants) | 18 | 19
hr*nmol/L
  Metabolite 1 (M1): number analyzed (Participants) | 18 | 18
  Metabolite 1 (M1) | 10550.8 (17276.38) | 15776.1 (29461.34)
  Metabolite 2 (M2) | 5880.6 (3404.27) | 5081.6 (3334.41)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to 30 days after the last dose of study drug (up to 12 months)
Population: Safety Population is defined as all participants who received at least 1 dose of any study drug and were used for all safety analyses. Although there were 2 parts to the study, however, data for adverse events was not collected separately for each part.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
Number analyzed (Participants) | 24
Participants
  AEs | 24
  SAEs | 12

11. Secondary Outcome: Number of Participants With Abnormal Laboratory Values Reported as AEs
Description: Standard safety laboratory tests included Chemistry and Hematology. Abnormal laboratory values that led to discontinuation or delay in treatment, dose modification, therapeutic intervention, or were considered by the investigator to be a clinically significant change from baseline were reported as AEs.
Time Frame: First dose of study drug to 30 days after the last dose of study drug (up to 12 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
Number analyzed (Participants) | 24
Participants
  Hypokalemia | 3
  Elevated blood creatinine | 3
  Increased international normalized ratio | 2
  Hypercalcemia | 1
  Hypomagnesemia | 1
  Hypoalbuminemia | 1
  Decreased blood potassium | 1
  Decreased blood sodium | 1
  Elevated blood alkaline phosphatase | 1
  Anemia | 5
  Neutropenia | 4
  Leukopenia | 2
  Thrombocytopenia | 2
  Decreased lymphocyte count | 2
  Decreased white blood cell count | 1
  Decreased platelet count | 1

12. Secondary Outcome: Number of Participants With Clinically Significant Change in Weight Reported as AEs
Description: Change relative to baseline in participant's weight measured throughout study.
Time Frame: First dose of study drug to 30 days after the last dose of study drug (up to 12 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
Number analyzed (Participants) | 24
Participants | 2

13. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Sign Reported as AEs
Description: Vital signs will include body temperature (oral), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Time Frame: First dose of study drug to 30 days after the last dose of study drug (up to 12 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib Without Itraconazole
Number analyzed (Participants) | 24
Participants
  Pyrexia | 3
  Palpitations | 2
  Tachycardia | 1

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 30 days after the last dose of study drug (up to 12 months)
Description: Although there were 2 parts to the study, however, data for adverse events was not collected separately for each part.
Arm/Group | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 12/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg (N=24)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Gait disturbance (General disorders) | 1
Disease progression (General disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment-emergent death occurred during treatment and is not related with study drug.
Haemorrhage intracranial (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Alisertib 30 mg+Itraconazole; Part B: Alisertib 50 mg (N=24)
Nausea (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 6
Gait disturbance (General disorders) | 3
Pyrexia (General disorders) | 3
Chills (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 5
Dysarthria (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 3
Confusional state (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 3
International normalised ratio increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Fall (Injury, poisoning and procedural complications) | 4
Palpitations (Cardiac disorders) | 3
Vision blurred (Eye disorders) | 2
Micturition urgency (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.